CLINICAL TRIAL: NCT03272750
Title: Controlled, Randomized, Double Blind Study, for the Evaluation of Tolerance and Trichological Efficacy of a Food Supplement: Bioscalin® New Formulation Versus Reference Formulation Currently on the Market and Placebo
Brief Title: Evaluation of Tolerance and Trichological Efficacy of a Food Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Dermatologist, Principal Investigator, Derming SRL
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E1416
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Telogen Effluvium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bioscalin® new formulation with Galeopsis Segetum (Experimental): 2 placebo capsules + 1 Bioscalin with Galeopsis Segetum table
  Interventions: Dietary Supplement: Bioscalin® new formulation with Galeopsis Segetum
- REFERENCE PRODUCT (Active Comparator): 2 reference product capsules + 1 placebo tablet
  Interventions: Dietary Supplement: Reference product
- PLACEBO (Placebo Comparator): 2 placebo capsules + 1 placebo tablet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bioscalin® new formulation with Galeopsis Segetum — Total duration of the study was 4 months; each subject, took by mouth two capsules/die of placebo at breakfast and one tablet/die of study product at lunch for the first 3 months of the trial.
  Arms: Bioscalin® new formulation with Galeopsis Segetum
Dietary Supplement: Reference product — Total duration of the study was 4 months; each subject, took by mouth two capsules/die of reference product at breakfast and one tablet/die of placebo at lunch for the first 3 months of the trial.
  Arms: REFERENCE PRODUCT
Dietary Supplement: Placebo — Total duration of the study was 4 months; each subject, took by mouth two capsules/die of placebo at breakfast and one tablet/die of placebo at lunch for the first 3 months of the trial.
  Arms: PLACEBO

SUMMARY:
Controlled, randomized, double blind study, for the evaluation of tolerance and trichological efficacy of a food supplement: Bioscalin® new formulation versus reference formulation currently on the market and placebo

DETAILED DESCRIPTION:
Aim of the study was to evaluate clinically and by non-invasive instrumental measurements the trichological activity of a food supplement taken for 3 months by subjects of both sexes, aged between 18-60 years, affected by telogen effluvium, with a percentage of hair in anagen phase < 75%.

In particular the study foresaw the evaluation of the trichological activity of the Bioscalin® new formulation with Galeopsis Segetum in comparison to a reference product currently on the market and to placebo.

It was also aim of this study to evaluate treatment tolerance.

ELIGIBILITY:
Inclusion Criteria:

* both sexes;
* age range 18-60 years old;
* with telogen effluvium and a percentage of anagen ratio at inclusion < 75%;
* no-smokers;
* accepting to follow the instruction received by the investigator;
* disposable and able to return to the study centre at the established times;
* accepting to not change their habits regarding food, physical activity, hair and scalp cleansing;
* accepting to not receive any drugs/cosmetics treatment able to interfere with the study results;
* no participation in a similar study actually or during the previous 6 months;
* accepting to sign the Informed consent form.

Exclusion Criteria:

* Pregnancy (for female subjects);
* lactation (for female subjects);
* subjects not in menopause who does not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test during the basal visit, after 2 (T2) and 3 (T3) month-treatment;
* change in the normal habits regarding food, physical activity, physical activity, hair and scalp cleansing during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit). The product contains gluten (aroma of grain), then all subjects with celiac disease or gluten intolerance should be excluded.
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study actually or during the previous 6 months.
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* clinical and significant skin condition on the test area (e.g. active eczema, dermatitis, psoriasis etc.).
* Diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy
* anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* assumption of drugs able to influence the test results in the investigator opinion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the percentage of hair in anagen phase | Basal visit (T0),1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4).
  Percentage of hair in anagen phase (anagen hair grow > 0,3 mm/die ) was calculate by TrichoScan software on the microscopic images (with 20X magnification) captured with FotoFinderDermoscope.
Change from baseline of the hair density | Basal visit (T0),1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4).
  Hair density (hair number/cm2) was calculate by TrichoScan software on the microscopic images (with 20X magnification) captured with FotoFinderDermoscope.
Change from baseline of the percentage of vellus hair | Basal visit (T0),1 month (T1), 2 months (T2), 3 months (T3), 4 months (T4).
  Percentage of vellus hair (vellus hair has a diameter <0.04 mm)was calculate by TrichoScan software on the microscopic images (with 20X magnification) captured with FotoFinderDermoscope.

SECONDARY OUTCOMES:
Hair parting test | Basal visit (T0), after 1 (T1), 2 (T2) and 3 (T3) month-treatment and a follow-up visit 1 month after the last food supplement assumption (T4 months).
  Evaluation of hair thickening
Videodermatoscopy | Basal visit (T0), after 1 (T1), 2 (T2) and 3 (T3) month-treatment and a follow-up visit 1 month after the last food supplement assumption (T4 months).
  Evaluation to visualize any morphological alteration/variation of the hair often imperceptible to the naked eye
Pull test | Basal visit (T0), after 1 (T1), 2 (T2) and 3 (T3) month-treatment and a follow-up visit 1 month after the last food supplement assumption (T4 months).
  Evaluation of tensile strength of the hair
Sebometry | Basal visit (T0), after 1 (T1), 2 (T2) and 3 (T3) month-treatment and a follow-up visit 1 month after the last food supplement assumption (T4 months).
  Measurement of surface lipid level